CLINICAL TRIAL: NCT04408690
Title: A Pilot Study to Investigate the Feasibility of Conducting a Randomized Controlled Trial That Compares Immediate Versus Optional Delayed Surgical Repair for Treatment of Acute Anterior Cruciate Ligament Injury
Brief Title: Feasibility of a RCT That Compares Immediate Versus Optional Delayed Surgical Repair After ACL Injury
Acronym: IODA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Federaal Kenniscentrum voor de Gezondheidszorg (Unknown); Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S62004
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation and optional delayed ACL reconstruction (Experimental)
  Interventions: Other: Rehabilitation; Procedure: Optional delayed anterior cruciate ligament reconstruction
- Immediate ACL reconstruction + rehabilitation (Active Comparator)
  Interventions: Procedure: Immediate anterior cruciate ligament reconstruction; Other: Rehabilitation

INTERVENTIONS:
Procedure: Immediate anterior cruciate ligament reconstruction — No guidelines on type of ACL reconstruction will be imposed to keep the trial pragmatic. The decision of graft type and surgery technique is a clinical decision made by the orthopaedic surgeons of the participating centra.
  This surgery will be performed within 12 weeks after the ACL injury.
  Arms: Immediate ACL reconstruction + rehabilitation
Other: Rehabilitation — All patients complete rehabilitation under supervision of their own physiotherapist. The investigators will provide some guidelines and criteria, but it is the physiotherapist's choice how to implement these guidelines in clinical practice.
Procedure: Optional delayed anterior cruciate ligament reconstruction — If a patient complains about persistent symptomatic instability of the knee or the inability to progress in rehabilitation, delayed surgery can be considered. ACL insufficiency induced instability in combination with a positive pivot shift and an additional MRI are needed to confirm the cause of instability.
  This surgery will not be performed within the first 12 weeks after the ACL injury.
  Arms: Rehabilitation and optional delayed ACL reconstruction

SUMMARY:
Currently, most patients with an anterior cruciate ligament (ACL) injury undergo surgery. There is a general belief that surgical reconstruction is necessary to return to sport safely and to limit premature knee osteoarthrosis or additional meniscal damage. However, there is unsufficient scientific evidence for this belief. Moreover, several studies show that a reconstruction does not guarantee successful return to sports or the prevention of osteoarthritis or meniscal injuries at all. Therefore, an immediate surgery after an ACL injury is more and more questioned. The only qualitative RCT that exists (KANON trial) could not demonstrate that an immediate reconstruction is an added value (in terms of symptoms, knee function, activity level, osteoarthritis or incidental meniscal damage) compared to a conservative approach consisting of progressive rehabilitation and delayed surgery if there was persistent knee instability.

In a future multicenter RCT the investigators want to 1) verify these results and 2) search for predictors that predict which patients from the conservative group do well without delayed surgery. This information is invaluable to physicians as it allows them to decide which treatment is best for the patient.

Before performing a large, adequately-powered RCT that compares both treatment options, the investigators will run a pilot study that assesses the feasibility to recruit ACL patients for such RCT. This seems necessary, as many patients still believe that timely surgery is a prerequisite for restoring knee function, for returning to sports and for preventing cartilage degeneration. These preferences for surgery might affect recruitment and adherence to the protocol. Therefore, a pilot study will performed that demonstrates whether a large RCT is feasible with regard to 1) participant recruitment, 2) adherence to the treatment arm they were allocated to and 3) protocol feasibility. The findings of this pilot study will help deciding about progressing to a future definitive RCT.

ELIGIBILITY:
Inclusion Criteria:

* Rotational trauma to a previously uninjured knee within the preceding 4 weeks
* Medical diagnosis of ACL insufficiency including MRI (both partial and complete ruptures)
* Minimum of 18 years

Exclusion Criteria:

* Patient has history of a previous ACL injury or knee surgery to the index knee.
* Indication for acute surgery because of related injuries to the knee
* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Female who is pregnant. Since MRI assessment cannot be performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Feasibility to recruit patients: Number of eligible patients that sign the informed consent | 4 months after first patient in
  Number of eligible patients that sign the informed consent

SECONDARY OUTCOMES:
Feasibility of the protocol: Number of patients that complete all assessments | When 5 patients per site have completed the 3 month follow-up visit
  Number of patients that complete all assessments (at baseline and 3 month follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Koen Peers, MD, PhD, Principal Investigator — UZ Leuven
Locations (2):
- Belgium (2):
  - UZ Leuven, Leuven
  - CHU Liège, Liège

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ghafelzadeh Ahwaz F, Smeets A, Bogaerts S, Berger P, Peers K. The feasibility of conducting a randomized controlled trial that compares immediate versus optional delayed surgical repair for treatment of acute Anterior cruciate ligament injury-results of the IODA pilot trial. Pilot Feasibility Stud. 2025 May 8;11(1):63. doi: 10.1186/s40814-025-01652-2. PMID 40340976
- [Derived] Smeets A, Ghafelzadeh Ahwaz F, Bogaerts S, De Groef A, Berger P, Kaux JF, Daniel C, Croisier JL, Delvaux F, Laenen A, Staes F, Peers K. Pilot study to investigate the feasibility of conducting a randomised controlled trial that compares Immediate versus Optional Delayed surgical repair for treatment of acute Anterior cruciate ligament injury: IODA pilot trial. BMJ Open. 2022 Mar 11;12(3):e055349. doi: 10.1136/bmjopen-2021-055349. PMID 35277406